CLINICAL TRIAL: NCT06666192
Title: A Multi-Level Intervention for Improving Screening Rates of Breast, Cervical and Colorectal Cancer in Women in Low-Income Communities
Brief Title: The Ohio State University (OSU) SCREEN Community Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: OSU-23400; NCI-2024-07400 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma; Cervical Carcinoma; Colorectal Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms | interventions — Mass Screening; Early Intervention, Educational; Educational Status; Methods; Focus Groups; Delivery of Health Care; Health Promotion; Risk Assessment; Interviews as Topic; Community-Institutional Relations; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Phase I, Planning Phase (MLI material, focus group, interview) (Other): Providers and community members review MLI materials and participate in focus groups and interviews to discuss challenges to being screened, what community members know about cancer and screening and what should be included in a program to increase screening over 30-60 minutes on study. A clinic champion will be identified during the interview to lead, advise, and oversee the implementation of the MLI at their clinic location.
  Interventions: Behavioral: Focus Group; Other: Informational Intervention; Other: Interview
- Phase II, Arm I (Health Clinics) (Active Comparator): The clinic champion coordinates planning sessions, staff training, and overall implementation and planning for the MLI within each health clinic. Health clinics may integrate new activities into usual clinic processes such as the use of the EHR to identify age-eligible patients in need of breast, cervical and/or CRC screening, reminder systems built into the EHR that can be sent to both providers and patients for screening and follow-up, and EHR information alerts for providers about patients who have positive FITs or a positive Pap test or mammogram on study. Additionally, health clinics may incorporate risk assessments (via paper or within the EHR) for all patients eligible for breast, cervical and/or CRC screening, promote screening via web-based or health portal messaging, promote annual wellness visits (during which screening should be discussed), and offer incentives for completing needed cancer screening on study.
  Interventions: Other: Health Care Delivery; Other: Health Promotion; Behavioral: Health Risk Assessment; Procedure: Implementation; Behavioral: Patient Navigation
- Phase II, Arm II (Health Care Providers) (Active Comparator): Providers participate in educational sessions that include self-administered pre-test surveys and discussions that assess screening knowledge, beliefs, attitudes, and practices, over one hour on study. Providers may also undergo coaching calls and one-on-one discussions to help tailor information and its delivery to the needs of providers and practices and are taught how to use clinic-based scheduling and reminder systems to help facilitate screening and follow-up actions.
  Interventions: Other: Discussion; Other: Educational Activity; Other: Health Care Delivery; Other: Health Promotion and Education; Other: Survey Administration
- Phase II, Arm III (Patients) (Active Comparator): Patients receive educational materials about screening and screening recommendations via mail and during in-person visits, and a web link for the developed small media website on study. Patients participate in discussions about screening and are offered any test for which they are not up to date and appropriate follow-up is conducted by designated staff on study. Patients who choose to undergo testing and receive a positive result receive a letter from the clinic and a call from the designated clinic staff member on study.
  Interventions: Other: Cancer Screening; Other: Discussion; Other: Educational Intervention; Other: Internet-Based Intervention
- Phase II, Arm IV (Community) (Active Comparator): Community receive educational materials (e.g., posters) and outreach activities to promote screening (e.g., health fairs, farmers' markets, inflatable colon tours, community seminars) and receive access to a CHW for one-on-one education about screening on study.
  Interventions: Other: Discussion; Other: Educational Intervention; Behavioral: Outreach; Behavioral: Patient Navigation
- Phase III and IV, Arm V (MLI Early Wave) (Experimental): Participating clinics and communities participate in the MLI early (years 2-3) for up to 30 months.
  Interventions: Other: Health Promotion and Education
- Phase III and IV, Arm VI (MLI Delayed Wave) (Experimental): Participating clinics and communities participate in the MLI 12 months later (years 3-4) for at least 12 months.
  Interventions: Other: Health Promotion and Education

INTERVENTIONS:
Other: Cancer Screening — Undergo cancer screening
  Other Names: Cancer Screening for Patients; Early Cancer Detection; Screening; Screening of Cancer
  Arms: Phase II, Arm III (Patients)
Other: Discussion — Participate in discussions
  Other Names: Discuss
  Arms: Phase II, Arm II (Health Care Providers); Phase II, Arm III (Patients); Phase II, Arm IV (Community)
Other: Educational Activity — Receive coaching calls
  Arms: Phase II, Arm II (Health Care Providers)
Other: Educational Intervention — Receive educational materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Phase II, Arm III (Patients); Phase II, Arm IV (Community)
Behavioral: Focus Group — Participate in focus group
  Arms: Phase I, Planning Phase (MLI material, focus group, interview)
Other: Health Care Delivery — Integrate new activities into usual clinic processes
  Other Names: Care Delivery; Health Services Delivery, Other; Healthcare Delivery
  Arms: Phase II, Arm I (Health Clinics); Phase II, Arm II (Health Care Providers)
Other: Health Promotion — Promote screening and wellness visits
  Other Names: Health Promotion (Salutogenesis); Health Promotion and Wellness; Mindfulness Health Promotion; Salutogenesis
  Arms: Phase II, Arm I (Health Clinics)
Other: Health Promotion and Education — Participate in educational sessions
  Arms: Phase II, Arm II (Health Care Providers)
Other: Health Promotion and Education — Participate in early wave MLI
  Arms: Phase III and IV, Arm V (MLI Early Wave)
Other: Health Promotion and Education — Participate in late wave MLI
  Arms: Phase III and IV, Arm VI (MLI Delayed Wave)
Behavioral: Health Risk Assessment — Incorporate risk assessments
  Other Names: Risk Assessment
  Arms: Phase II, Arm I (Health Clinics)
Procedure: Implementation — Implement MLI
  Arms: Phase II, Arm I (Health Clinics)
Other: Informational Intervention — Review MLI materials
  Arms: Phase I, Planning Phase (MLI material, focus group, interview)
Other: Internet-Based Intervention — Receive educational online materials
  Arms: Phase II, Arm III (Patients)
Other: Interview — Participate in interview
  Arms: Phase I, Planning Phase (MLI material, focus group, interview)
Behavioral: Outreach — Receive outreach activities
  Other Names: Outreach Strategy
  Arms: Phase II, Arm IV (Community)
Behavioral: Patient Navigation — Receive access to CHW
  Other Names: Patient Navigator Program
  Arms: Phase II, Arm I (Health Clinics); Phase II, Arm IV (Community)
Other: Survey Administration — Ancillary studies
  Arms: Phase II, Arm II (Health Care Providers)

SUMMARY:
This clinical trial develops and tests how well a multi-level intervention (MLI), The Ohio State University (OSU) SCREEN Community Program, works to increase screening and follow-up for breast, cervical and colorectal (CRC) cancer among low-income and un/underinsured female residents in three counties in Central Ohio. In Ohio, incidence and mortality rates for breast, cervical and CRC are higher than or similar to the national average; in addition, underserved populations - minority, rural and low-income women - have higher rates of these cancers. Screening can detect precancerous colorectal and cervical lesions and other early-stage cancers when treatment is less intensive and more successful and is known to reduce mortality rates for breast, cervical, and CRC, however many of these women lack access to health care and screenings. This MLI includes clinic-based components, such as patient education, as well as community-based strategies, such as media programs and training health workers, that can increase rates of guideline-recommended breast, cervical and CRC screening and follow-ups in underserved populations. The OSU SCREEN Community Program may be an effective way to improve breast, cervical and CRC screenings among underserved women in Ohio.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Understand local factors and context relevant to breast, cervical and CRC screening and follow-up (including referral-to-care) and develop an MLI planning and implementation pathway for use by partner health centers and communities (Year 1).

II. Pilot test and further refine the MLI planning and implementation process in one clinic (Years 1 & 2).

III. Test the final MLI planning and implementation process in a group randomized, delayed intervention trial to assess the impact of the customized MLI on increasing rates of guideline recommended breast, cervical and CRC screening and follow-up for abnormal tests (Years 2, 3 and 4).

IV. Assess sustainability of the MLI (Years 4 and 5).

OUTLINE:

PHASE I (PLANNING): Providers and community members review MLI materials and participate in focus groups and interviews to discuss challenges to being screened, what community members know about cancer and screening and what should be included in a program to increase screening over 30-60 minutes on study. A clinic champion will be identified during the interview to lead, advise, and oversee the implementation of the MLI at their clinic location.

PHASE II (PILOT): Participants are assigned to 1 of 4 arms.

ARM I (HEALTH CLINICS): The clinic champion coordinates planning sessions, staff training, and overall implementation and planning for the MLI within each health clinic. Health clinics may integrate new activities into usual clinic processes such as the use of the electronic health record (EHR) to identify age-eligible patients in need of breast, cervical and/or CRC screening, reminder systems built into the EHR that can be sent to both providers and patients for screening and follow-up, and EHR information alerts for providers about patients who have positive fecal immunochemical test (FITs) or a positive Pap test or mammogram on study. Additionally, health clinics may incorporate risk assessments (via paper or within the EHR) for all patients eligible for breast, cervical and/or CRC screening, promote screening via web-based or health portal messaging, promote annual wellness visits (during which screening should be discussed), and offer incentives for completing needed cancer screening on study.

ARM II (HEALTH CARE PROVIDERS): Providers participate in educational sessions that include self-administered pre-test surveys and discussions that assess screening knowledge, beliefs, attitudes, and practices, over one hour on study. Providers may also undergo coaching calls and one-on-one discussions to help tailor information and its delivery to the needs of providers and practices and are taught how to use clinic-based scheduling and reminder systems to help facilitate screening and follow-up actions.

ARM III (PATIENTS): Patients receive educational materials about screening and screening recommendations via mail and during in-person visits, and a web link for the developed small media website on study. Patients participate in discussions about screening and are offered any test for which they are not up to date and appropriate follow-up is conducted by designated staff on study. Patients who choose to undergo testing and receive a positive result receive a letter from the clinic and a call from the designated clinic staff member on study.

ARM IV (COMMUNITY): Communities receive educational materials (e.g., posters) and outreach activities to promote screening (e.g., health fairs, farmers' markets, inflatable colon tours, community seminars) and receive access to a community health worker (CHW) for one-on-one education about screening on study.

PHASE III and IV: Participating clinics and surrounding communities are randomized to 1 of 2 arms.

ARM V (EARLY INTERVENTION WAVE): Participating clinics and communities participate in the MLI early (years 2-3) for up to 30 months.

ARM VI (DELAYED INTERVENTION WAVE): Participating clinics and communities participate in the MLI 12 months later (years 3-4) for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Level 1 is the health clinics (Helping Hands [pilot]; 6 Lower Lights clinics). Clinics are eligible if they provide preventive health care to residents of the targeted census tracts.
* Level 2 focuses on health care providers (physicians, nurses, physician assistants [PA]/nurse practitioners [NPs]) and office staff practicing at participating clinics who are involved in the screening and/or screening referral process (determined by individual clinical sites) and can speak, read, and write English
* Patients (Level 3) are the recipients of health care and screening interventional strategies implemented by clinics and providers.
* Level 4 is the community to include residents in targeted census tracts around each clinic.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2067 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Up to date (UTD) status for all three screenings (Early Intervention Wave) | At baseline and at the end of the Implementation Phase (up to 4 years)
  Will be assessed by the difference in proportions of being UTD with all age-appropriate screening tests using electronic health record (EHR) data. Rates will be examined by age, race/ethnicity, residence, payer status, provider, time since last visit, and rates of other cancer screening. Repeated measure Generalized Estimating Equations (GEE) models with compound symmetry correlation structure and robust variance will be used to compare change between the early and delayed intervention groups adjusting for baseline UTD screening rates of the targeted communities. Adjustment for baseline UTD screening rates and rates of follow up for abnormal test will control for any differences by intervention group due to chance and will increase power by decreasing the standard error of the treatment effect. To account for differences in number of respondents across targeted communities, GEE models will be weighted using an approach described by Johnson et al.
Status of follow-up for abnormal tests (Early Intervention Wave) | At baseline and at the end of the Implementation Phase (up to 4 years)
  Will be assessed by the difference in follow-up rates for abnormal tests using EHR data. GEE models with compound symmetry correlation structure and robust variance will be used to compare change between the early and delayed intervention groups adjusting for baseline UTD screening rates of the targeted communities. Adjustment for baseline UTD screening rates and rates of follow up for abnormal test will control for any differences by intervention group due to chance and will increase power by decreasing the standard error of the treatment effect. To account for differences in number of respondents across targeted communities, GEE models will be weighted using an approach described by Johnson et al.

SECONDARY OUTCOMES:
UTD screening status for all three cancers and follow up rates for abnormal tests | At the end of early intervention (up to 2.5 years)
  Will be assessed among age-appropriate residents of targeted census tracts. The individual-level UTD status pre- and post-intervention will be obtained from cross-sectional surveys, and it will be defined based on the age-specific United States Preventive Services Task Force Cancer Screening Guidelines screening recommendations for each cancer. A two-level hierarchical mixed-effects logistic regression model will be used to compare the UTD odds between the early and delayed intervention groups. In this two-level design, participants are the level one unit while the clinic areas are the level two unit of analysis, with all subjects in each cluster receiving either the early or delayed intervention. This design will allow to examine the effectiveness of the multi-level intervention at the individual- and cluster levels.

CONTACTS AND LOCATIONS:
Overall Officials: Electra D Paskett, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu